CLINICAL TRIAL: NCT04903262
Title: Strategy of Ultra-Protective Lung Ventilation With Extracorporeal CO2 Removal for New-Onset Moderate ARDS: A Prospective Multicenter Randomized Clinical Trial
Brief Title: Ultra-Protective Lung Ventilation With Extracorporeal CO2 Removal for Moderate ARDS
Acronym: SUPERNOVA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bologna (Other)
Collaborators: Getinge Group (Other)
Responsible Party: Principal Investigator, V. Marco Ranieri, Full Professor, University of Bari Aldo Moro
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SUPERNOVA
Record Dates: First submitted 2021-05-21; First posted 2021-05-26 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ECCO2R (Experimental): Patients will be initially treated with "standardized ventilation": volume assist/control, VT = 6 mL/kg PBW; insp. flow 50-70 L/min, I:E ratio 1:1 to 1:3; RR 20-35 bpm; PEEP according to "low PEEP/ high FiO2" table. Goals: PaO2 55-80 mmHg or SpO2 88-95%; arterial pH: 7.30-7.45.
  ECCO2R initiated during "standardized ventilation" with blood flow between 1000 and 1500 mL/min. Anticoagulation with unfractionated heparin to a target aPTT of 1.5-2.0x baseline. Target: maintain PaCO2 at baseline ± 20%.
  VT initially reduced to 5 mL/kg. Sweep gas initiated and VT decreased to 4.5 then 4 mL/kg; PEEP adjusted to maintain same mean airway pressure as during "standardized ventilation", provided that Pplat ≤ 25 cmH2O.
  Respiratory rate decreased to 8 bpm. If PaCO2 > 75 mmHg and/or pH < 7.2, despite respiratory rate of 35/min and optimized ECCO2R, VT will be increased to the last previously tolerated VT.
  Recommendation: 2 daily lung recruitment maneuvers (as per clinical practice in each center).
  Interventions: Procedure: Ultraprotective ventilation with Extracorporeal CO2 removal
- Standard of care (Active Comparator): Patients will be treated with "standardized ventilation": volume assist/control, VT = 6 mL/kg PBW; insp. flow 50-70 L/min, I:E ratio 1:1 to 1:3; RR 20-35 bpm; PEEP according to "low PEEP/ high FiO2" table. Goals: PaO2 55-80 mmHg or SpO2 88-95%; arterial pH: 7.30-7.45.
  Recommendation: 2 daily lung recruitment maneuvers (as per clinical practice in each center).
  Interventions: Procedure: Conventional protective ventilation

INTERVENTIONS:
Procedure: Ultraprotective ventilation with Extracorporeal CO2 removal — HLS5.0 Cardiohelp® (Getinge Cardiopulmonary Care, Rastatt, Germany): 1.3 m² polymethylpentene hollow fiber membrane oxygenator. The extracorporeal blood flow is in the range of 1000 to 1500 mL/min. Sweep gas (air or oxygen) is drawn through the hollow fibers by a vacuum pump, creating a diffusion gradient for gas exchange across the membrane.
  Arms: ECCO2R
Procedure: Conventional protective ventilation — Conventional lung protective mechanical ventilation, as described in the arm description ("standardized ventilation")
  Arms: Standard of care

SUMMARY:
Acute respiratory distress syndrome (ARDS) accounts for 10% of all ICU admissions and for 23% of patients requiring mechanical ventilation (MV). Its hospital mortality remains high, ranging from 34% in mild forms up to 46% in severe cases. Positive pressure MV remains the cornerstone of management, but at the same time it can contribute to worsening and maintenance of the lung injury when excessive stress and strain is applied to the lung parenchima (so-called ventilator-induced lung injury, VILI). VILI significantly contributes to the morbidity and mortality of ARDS patients, and it has been clearly demonstrated that protective (low-volume, low-pressure) MV settings are associated with a significant survival benefit. Unfortunately, in a certain proportion of ARDS cases, it is difficult to preserve acceptable gas exchange while maintaining protective ventilation settings, due to a high ventilatory load. In these cases, extracorporeal CO2 removal (ECCO2R) can be applied to grant the application of protective or even ultra-protective mechanical ventilation settings.

The main outcome of this multicenter, prospective, randomized, comparative open trial is to determine whether early ECCO2R allowing ultraprotective mechanical ventilation improves the outcomes of patients with moderate ARDS.

DETAILED DESCRIPTION:
Acute respiratory distress syndrome (ARDS) represents a form of lung injury that occurs in response to various predisposing events, characterized by inflammation, increased pulmonary vascular permeability and loss of aerated lung tissue. The diagnosis of ARDS is based on severe hypoxemia and bilateral radiographic opacities occurring within 7 days of a known clinical insult or worsening respiratory symptoms. Central to the pathophysiology of ARDS is the presence of fibrin-rich exudates (hyaline membranes) due to activation of coagulation and inhibition of fibrinolysis. ARDS accounts for 10 % of all ICU admissions and for 23% of patients requiring mechanical ventilation (MV). Hospital mortality of ARDS patients remains high, ranging from 34% with mild ARDS, up to 46% with severe ARDS. Notably, severe and critical forms of coronavirus disease 2019 (COVID-19) are almost invariably associated with ARDS.

Ventilator Induced Lung Injury (VILI) MV is a lifesaving form of support for patients with ARDS since it decreases the oxygen cost of breathing, improves gas exchange and provides time for resolution of the underlying etiology of ARDS. However, it has been consistently shown that MV may contribute to ventilator-induced lung injury (VILI) characterized by progression of pulmonary damage, worsening of the pulmonary inflammatory process, increased alveolar-capillary permeability and therefore leading to the translocation of inflammatory mediators from the lungs into the systemic circulation with consequent failure of distal organs (biotrauma). A randomized clinical trial showed that ventilating ARDS patients with a tidal volume (VT) of 6 ml/kg (calculated from predicted body weight, PBW), and with a maximum end-inspiratory plateau pressure (PPLAT) of 30 cmH2O decreased mortality from 40 % (seen in the conventional arm treated with a VT of 12 ml/kg PBW) to 31%. Recently, Amato and coworkers showed that the delta pressure (∆P), i.e. the difference between PPLAT and positive end-expiratory pressure (PEEP) (∆P = PPLAT -PEEP) ≤ 14 cmH2O was strongly associated with survival, demonstrating that interventions to obtain protective ventilatory settings (reductions in VT or increases in PEEP) were beneficial only if associated with decreases in ΔP.

Extra-corporeal CO2 Removal (ECCO2-R) The use extracorporeal support to remove carbon dioxide (CO2) to permit the use of low volume/low pressure ventilation with minimal impact on PaCO2 was proposed in 1977. It was suggested that applying low VT and low peak inspiratory pressures ("lung rest") at a low respiratory rate could minimize damage to the compromised lungs. With this technique, oxygenation and removal of carbon dioxide were dissociated: oxygenation occurred predominantly through the lungs, and a variable portion of the carbon dioxide was removed through an artificial lung (extracorporeal CO2removal: ECCO2-R). The key potential advantage to this approach over extracorporeal membrane oxygenation (ECMO) is the use of lower blood flow through the extracorporeal circuit potentially with fewer side effects. Low VT ventilation (3-4 ml/kg of PBW) was associated with a significant decrease in inflammatory markers when compared with standard low volume, low pressure ventilation. Furthermore, the resulting hypercapnia was easily controlled by ECCO2-R. A randomized clinical trial showed that VT of 3 ml/kg of PBW was easy and safe to be implemented with extracorporeal CO2-removal. Clinical outcome, evaluated as days free from mechanical ventilation through day 28, significantly improved in ECCO2R patients compared to control, when analyzing patients with PaO2/FiO2<150.

A multicenter study designed to assess safety and feasibility of ECCO2R in ARDS showed that more than 80% of patients with moderate ARDS could achieve ultra-protective ventilation goals by using ECCO2R. The incidence of severe adverse events related to ECCO2R was low (~2%). Efficacy and safety of ECCO2R A was higher for devices that used blood flow rates in the range of 1000-1500 ml/min. A post-hoc analysis showed that restricting enrollment to patients with compliance of the respiratory system ≤ 40 ml/cmH2O and decrease in ∆P ≥ 5 cmH2O would increase predicted benefit in terms of clinical outcomes in a randomized clinical trial of VT of 3 ml/kg of PBW with ECCO2R (enrichment strategy). Moreover, recent data show that there is no safe upper limit for PPLAT or ΔP, consistent with the fact that since the mortality rate in ARDS patients with ΔP values ≤ 14 cmH2O is still as high as 20%. Patient outcomes may therefore be improved by aggressively lowering ventilatory variables such as VT, PPLAT, or ΔP as facilitated by ECCO2R devices that remove CO2. In addition, ECCO2R might further decrease VILI by allowing lower respiratory rates, which have been shown to be lung protective.

OBJECTIVE The objective of this multicenter, prospective, randomized, comparative open trial is to determine if early ECCO2R allowing ultraprotective mechanical ventilation (VT 4 ml/kg) improves the outcomes of patients with ARDS.

PROCEDURES

CONTROL GROUP

* Patients will be treated with the following conventional ventilator settings ("standardized ventilation"): mode of mechanical ventilation: volume assist/control; VT = 6 mL/kg (PBW); inspiratory flow will be set at 50-70 L/min resulting in an end-inspiratory pause of 0.2-0.5 sec, I:E ratio 1:1 to 1:3; set RR to 20-35 bpm; PEEP will be set according to the "lower PEEP/FiO2" table:
* PBW will be calculated according to the following formulae: PBW (Males) = 50 + 0.91 [height (cm)-152.4]; PBW (Females) = 45.5 + 0.91 height (cm)-152.4].
* Oxygenation Goal: PaO2 55-80 mmHg or SpO2 88-95%;
* Arterial pH Goal: 7.30-7.45.
* It is recommended to perform 2 daily lung recruitment maneuvers (as per standard clinical practice in each center).
* Patients may receive NMBA and continued as directed by the attending physician.
* Use heated humidifiers for gas humidification and minimize instrumental dead space.

TREATMENT GROUP

* Patients will be treated with the following conventional ventilator settings ("standardized ventilation"): mode of mechanical ventilation: constant flow, volume assist/control; VT = 6 mL/kg (PBW); inspiratory flow will be set at 50-70 L/min resulting in an end-inspiratory pause of 0.2-0.5 sec, I:E ratio 1:1 to 1:3; set RR to 20-35 bpm; PEEP will be set according to the "lower PEEP/FiO2" table:
* PBW will be calculated according to the following formulae: PBW (Males) = 50 + 0.91 [height (cm)-152.4]; PBW (Females) = 45.5 + 0.91 height (cm)-152.4].
* Oxygenation Goal: PaO2 55-80 mmHg or SpO2 88-95%;
* Arterial pH Goal: 7.30-7.45.
* Patients may receive NMBA and continued as directed by the attending physician.
* Use heated humidifiers for gas humidification and minimize instrumental dead space.
* ECCO2R will be initiated during "standardized ventilation".
* Catheterization for ECCO2R will be performed according to local institutional clinical practice. The ECCO2R circuit will be connected to the catheter and blood flow set between 1000 and 1500 mL/min. Initially, sweep gas flow through the ECCO2R device will be set at zero (0 LPM) such as to not initiate CO2 removal through the device. Anticoagulation will be maintained with unfractionated heparin to a target aPTT of 1.5 - 2.0x baseline. A bolus of 80 I.U./kg unfractionated heparin is suggested at the time of cannulation.
* The objective is to maintain PaCO2 at baseline value ± 20% of baseline settings obtained with a VT = 6 mL/kg provided that pH remains ≥ 7.30. End-tidal CO2 (EtCO2) will be monitored for safety purposes.
* REDUCTION OF VT: Following a run-in time (up to a maximum of 2 hours) with sweep gas flow at zero LPM, VT will be reduced gradually to 5 mL/kg. Sweep gas will be initiated and VT decreased to 4.5 then 4 mL/kg, and PEEP adjusted to maintain the same mean airway pressure as during standardized ventilation, provided that Pplat ≤ 25 cmH2O (i.e., if the PEEP level required to maintain mean airway pressure leads to a Pplat > 25 cmH2O, PEEP is then reduced until a Pplat ≤ 25 cmH2O).
* It is recommended to perform 2 daily lung recruitment maneuvers (as per standard clinical practice in each center).
* REDUCTION OF RESPIRATORY RATE: Respiratory rate will be progressively decreased to a minimum of 8 bpm and facilitated by increases in sweep gas flow; a constant I:E ratio will be maintained.
* If PaCO2 > 75 mmHg and/or pH < 7.2, despite respiratory rate of 35/min and optimized ECCO2R, VT will be increased to the last previously tolerated VT.
* CO2 removal will be performed using the following device, routinely used for clinical purposes in each site:
* HLS5.0 Cardiohelp® (Getinge Cardiopulmonary Care, Rastatt, Germany): 1.3 m² polymethylpentene hollow fiber membrane oxygenator will be used, combined with HLS sets (BIOLINE heparine-coating). The extracorporeal blood flow is in the range of 1000 to 1500 mL/min. Sweep gas (air or oxygen) is drawn through the hollow fibers by a vacuum pump, creating a diffusion gradient for gas exchange across the membrane.

INTERRUPTION OF TREATMENT According to group assignment, "standardized ventilation" or "ultra protective ventilation + ECCO2R" will be maintained for at least 72 hours; then, interruption trials according to protocol will be performed every 24 hours, until liberation from mechanical ventilation and ECCO2R. In the treatment group, patients will be always weaned first from ECCO2R and subsequently from mechanical ventilation.

Interruption trials will be performed after at least 72 hours of study enrollment if all the following criteria are met: 1) PaO2/FiO2 > 250 with PEEP 8-10 cmH2O and FiO2 <0.5; 2) values of both PEEP and FIO2 ≤ than values from previous day; 3) the patient is not receiving neuromuscular blocking agents; 4) the patient is exhibiting inspiratory efforts; 5) systolic arterial pressure ≥ 85 mmHg without vasopressor and/or inotropic support (≤ 5 mcg/kg/min dopamine or dobutamine will not be considered inotropic support in this context).

In the CONTROL group, in presence of all criteria 1-5, a spontaneous breathing trial will be conducted every 24 hours, until liberation from mechanical ventilation (see "weaning procedures" below).

In the TREATMENT group, in presence of all criteria 1-5, a zero-sweep gas trial will be conducted every 24 hours: sweep gas will be deactivated for 6 hours and then presence of all criteria 1-5 will be checked again; if still all present, ECCO2R will be removed and further weaning from mechanical ventilation will be conducted as in the control group.

RESCUE THERAPIES

* Refractory hypoxemia will be defined as PaO2 < 60 mm Hg for at least 1 hour while receiving an FIO2 of 1.0
* Refractory acidosis will be defined as pH ≤ 7.10 for at least 1 hour
* Refractory barotrauma will be defined as persistent pneumothorax with 2 chest tubes on the involved side or increasing subcutaneous or mediastinal emphysema with 2 chest tubes.

If refractory hypoxemia OR refractory acidosis OR refractory barotrauma occurs, the events surrounding this event(s) will be recorded and clinicians at their discretion may deviate from the assigned ventilation protocols and institute so-called rescue therapies, including: inhaled nitric oxide, prone position, extracorporeal membrane oxygenation (ECMO). The use of these therapies will be recorded in the study case report forms.

WEANING PROCEDURES

* A Spontaneous Breathing Trial (SBT) procedure and assessment for unassisted breathing will be performed: 30 - 120 minutes of spontaneous breathing with FIO2 < 0.5 using any of the following approaches: Pressure support (PS) < 5 cmH2O, PEEP < 5 cmH2O; CPAP < 5 cmH2O; T-piece; Tracheotomy mask
* Criteria to be met during the last 30 minutes of a SBT for reporting the SBT as "SUCCESSFUL": SpO2 ≥ 90% and / or PaO2 ≤ 60 mm Hg; Respiratory Rate ≤ 35 / min; pH ≥ 7.30; Absence of respiratory distress.
* If any of the above-mentioned criteria is not met, the SBT will be reported as "UNSUCCESSFUL" and previous ventilator settings or to PS greater than or equal to 10 cm H2O with PEEP and FIO2 at the previous settings will be initiated. The patient will be reassessed for weaning the following day.
* If the SBT is "SUCCESSFUL", ventilatory support will be removed.
* Patients will be reported as "VENTILATOR FREE" after two consecutive calendar days of "UNASSISTED BREATHING". "UNASSISTED BREATHING" will be defined as any of the following: Spontaneously breathing with face mask, nasal prong oxygen, or room air; T-tube breathing; Tracheostomy mask breathing; CPAP ≤ 5 without PS or IMV assistance; use of CPAP or BIPAP solely for sleep apnea management

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* On invasive mechanical ventilation for ≤ 96 hours
* Presence of all of the following conditions for ≤ 24 hours: 100 < PaO2/FiO2 ≤ 200 after 12 hours of "standardized ventilation" with PEEP ≥ 5; compliance of the respiratory system ≤ 0.5 ml/cmH2O per kg PBW; ventilatory ratio (VR) ≥ 1.5; bilateral opacities not fully explained by effusions, lobar/lung collapse, or nodules; respiratory failure not fully explained by cardiac failure or fluid overload

Exclusion Criteria:

* Pregnancy
* ARDS with PaO2/FiO2<100 or PaO2/FiO2>200 under standardized ventilation with PEEP ≥ 5 cmH2O
* Expected duration of mechanical ventilation < 48 hours
* Severe COPD
* Chronic respiratory insufficiency with home ventilation or oxygen therapy
* Currently receiving ECMO therapy
* Acute brain injury
* Severe liver insufficiency (Child-Pugh scores >7) or fulminant hepatic failure
* Heparin-induced thrombocytopenia
* Contraindication for systemic anticoagulation
* Platelet count <50,000/mm3
* Prothrombin time-international normalized ratio (INR) >1.5
* Patient moribund, decision to limit therapeutic interventions
* End-stage disease
* Unable to provide vascular access for ECCO2-R
* Acute coronary syndrome
* Actual body weight exceeding 1 kg per centimeter of height
* Burns > 40% total body surface
* Bone marrow transplantation within the last 1 year

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of ventilator-free days (VFDs) at 28 days after randomization. | 28 days
  VFD to-day 28 is defined as the number of days of unassisted breathing to day 28 after randomization, assuming a patient survives for at least two consecutive calendar days after initiating unassisted breathing and remains free of assisted breathing.

SECONDARY OUTCOMES:
28-day all-cause mortality | 28 days
  All patients will be classified as either "alive at Study Day 28" or, if dead, "dead at Study Day 28."
90-day all-cause mortality | 90 days
  All patients will be classified as either "alive at Study Day 90" or, if dead, "dead at Study Day 90".
Cumulative incidence of severe adverse events during 28 days after randomization | 28 days
  Device-related and/or patient-related severe adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Marco Ranieri, M.D., Study Chair — University of Bari; Antonio Pesenti, M.D., Study Chair — University of Milan
Locations (1):
- IRCCS AOUBO Policlinico di Sant'Orsola, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No